CLINICAL TRIAL: NCT07333885
Title: The Impact of Reducose® on Symptoms of Perimenopause and Glycemic Response: a Randomized Controlled Trial
Brief Title: Impact of Reducose® on Glycemic Response and Menopausal Symptoms in Perimenopausal Women (CALM-R)
Acronym: CALM-R
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Phynova Group Ltd (Industry)
Collaborators: People Science (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PYN-PS18-14914
Record Dates: First submitted 2025-12-19; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Glycemic Response; Menopause Symptoms
Keywords: Menopause

STUDY DESIGN:
Intervention Model Description: Parallel Assignment (two-arm RCT)
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This study is a randomized, double-blind, placebo-controlled trial. Participants, care providers, investigators, and outcomes assessors are blinded to intervention assignment. Study products are labeled as Product A or Product B, and the randomization code is maintained by the sponsor and only broken in the event of a serious adverse event.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reducose® Mulberry Leaf Extract (Experimental)
  Interventions: Dietary Supplement: Reducose® (Mulberry leaf extract)
- Matching Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Reducose® (Mulberry leaf extract) — Reducose® proprietary mulberry leaf extract, 250mg, 2/day with meals
  Arms: Reducose® Mulberry Leaf Extract
Dietary Supplement: Placebo — Placebo matching capsules, Microcrystalline Cellulose
  Arms: Matching Placebo

SUMMARY:
The purpose of this double-blind, randomized, placebo-controlled trial is to. evaluate daily Reducose® (mulberry leaf extract) supplementation taken with the two largest meals for 12 weeks on improving glycemic response and perimenopausal symptoms in women aged 40-60 years. Glycemic response is measured using Dexcom Stelo continuous glucose monitors during standardized test meals, and menopausal symptoms and sleep/quality-of-life outcomes are assessed using validated surveys administered through the Chloe app in a decentralized U.S. study.

ELIGIBILITY:
Inclusion Criteria:

* Participants assigned female at birth (aged 40-60 years) will be recruited for the study.
* Females ages 40-60 who are weight stable and with a self- reported Body Mass Index (BMI) between 18.5 to 35 kg/m2.
* Willing to maintain their existing dietary and physical activity patterns throughout the study period.
* Have received a medical physical screening (annual physical) within the last 12 months where blood markers for diabetes were taken and results were within the healthy range.
* Self-reported >40yrs in age and experiencing irregular periods.
* Willing and able to comply with the study protocol.
* Has given voluntary informed consent to participate in the study.
* Not currently using hormone replacement therapy (HRT) and/or >3months since their last hormone treatment.
* Experiencing menopause symptoms and meets the minimum score of 12/60 on the Greene Climacteric Scale (GCS).
* Own or have constant access to a smart phone and the apple or android app stores and are willing and able to download the Dexcom and Chloe apps and accept their respective privacy policies.
* Willing to practice a reliable method of non-hormonal contraception for the duration of the study.
* In good general health at the time of screening (Investigator discretion).
* Able to read, understand, and provide informed consent in English.
* Able to receive shipment of the product at an address within the United States.
* Able to complete study assessments over the course of up to 12 weeks.

Exclusion Criteria:

* Participants assigned male at birth.
* Aged > 60 or < 40 years.
* Pregnant or lactating.
* Body mass index (BMI) > 35kg/m2 or < 18.5kg/m2
* Fasting blood glucose >126mg/dL and/or HbA1c >6.5% reported in routine medical physical screening within the last 12-months.
* Known history of diabetes mellitus (Type I/II) or the use of antihyperglycemic drugs or insulin to treat diabetes and related conditions.
* Currently using hormone replacement therapy (HRT) or had hormone therapy in the last 3 months.
* Postmenopausal, experiencing amenorrhea for >12months.
* Underwent medically induced or surgical menopause.
* History of hysterectomy or full or partial oophorectomy.
* Any known food allergy or intolerance including mulberry extract.
* Medical condition(s) or medication(s) known to affect glucose regulation or appetite and/or influence digestion and absorption of nutrients, including thyroid conditions, active inflammatory bowel disease (Crohn's disease or ulcerative colitis) and incretin mimetics (GLP-1, Semaglutide, Dulagluetide, Tirzepatide, etc.)
* Previously undergone bariatric surgery.
* Use steroids, protease inhibitors, antipsychotics, antidepressants (including selective serotonin reuptake inhibitors and monoamine oxidase inhibitors) (all of which have effects on glucose metabolism and body fat distribution).
* Significant or untreated medical and/or psychiatric disorders including but not limited myocardial ischemia or infarction, unstable angina, uncontrolled hypertension, renal failure and serious renal diseases, undergoing dialysis, chronic active hepatitis, acute hepatitis, cirrhosis of liver, AIDS, malignancy or neurological disorders including epilepsy, recent cerebrovascular disease or recent traumatic brain injury.
* Alcohol intake above recommendations (>2 standard alcoholic drinks per day) or drug abuse or dependence within the past 6 months.
* Currently smoke tobacco and cannabis products (including vaping).
* Consuming extremely restrictive diet currently or within past 3 months.
* Weight has varied significantly (+/- 5 lbs) in the past 3 months.
* Cognitively impaired and/or who are unable to give informed consent.
* Taking daily medications or dietary supplements that have a significant effect on blood glucose control either as a primary function or side effect.
* Subject to a major medical, surgical or major depressive or psychiatric event requiring hospitalization within the preceding 3 months.
* Use of over the counter medications like Herbal Supplements: Black Cohosh, Dong Quai, Maca Root, Red Clover, Chaste Tree Berry (Vitex), Soy Isoflavones, Ashwagandha; OTC Non-Herbal Supplements: DHEA, Progesterone Cream (Bioidentical), Melatonin.
* Participation in any other clinical research trial within 30 days prior to randomization.
* Do not have a personal smartphone, internet access, or unwilling to download Chloe or use a Dexcom Continuous Glucose Monitoring Device.
* Are unlikely for any reason to be able to comply with the study protocol, do not provide informed consent, or considered unsuited for participation in the study by the Principal Investigator.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-12-12 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Glycemic response following test meal | Baseline and end-of-study test meals (Days 10, 14, and 98).
  Postprandial glycemic response measured as 0-120-minute incremental area under the curve (iAUC) from interstitial glucose readings captured by Dexcom Stelo CGM.

SECONDARY OUTCOMES:
Time to peak glucose (Tmax) following test meal | Days 10, 14, and 98.
  Time from start of test meal to maximum postprandial glucose level measured by CGM.
Peak glucose concentration (Cmax) following test meal | Days 10, 14, and 98.
  Maximum postprandial glucose level (mg/dL) measured by CGM.
Fasting blood glucose prior to test meals | Days 14 and 98.
  Fasting glucose level (mg/dL) obtained from CGM prior to test meals.
Mean Amplitude of Glycemic Excursions (MAGE) | Baseline (Days 7-14), Week 1 (Days 14-21), Week 11 (Days 85-92), Week 12 (Days 92-98).
  CGM-derived glycemic variability metric calculated over predefined baseline and follow-up windows.
Nighttime Gross Coefficient of Variation (%CV) | Baseline (Days 7-14), Week 1 (Days 14-21), Week 11 (Days 85-92), Week 12 (Days 92-98).
  CGM-derived nighttime glucose variability from 23:00-06:00.
Menopausal symptoms (Greene Climacteric Scale total score) | Screening/Day 0, Days 14, 42, 70, 98.
  Change in Greene Climacteric Scale (0-60) assessing vasomotor, somatic, psychological symptoms. The minimum possible score is 0 and the maximum possible score is 63 with a score of 21 indicating a woman is experiencing menopause-related symptom patterns. Direction of Improvement: Lower score indicates improvement.
Sleep disturbance (PROMIS Sleep Disturbance Short Form-6a) | Baseline (Day 5) and end of study (Day 98).
  Participant-reported sleep disturbance via validated PROMIS Sleep Disturbance-SF6a. For scoring, the raw score range of 8 (lowest possible) to 40 (highest possible). A score of 50 is average for sleep disturbance. Direction of Improvement: Higher score indicates improvement.
Quality of Life questionnaire | Baseline (Day 5) and end of study (Day 98).
  App-based questionnaires assessing perceived quality of life changes. Direction of Improvement: Higher score indicates improvement.
Product Experience Questionnaire | End of study (Day 98)
  Questionnaire for experience while taking product and use of Chloe App. Higher score indicates higher satisfaction with product and use of Chloe App,.

CONTACTS AND LOCATIONS:
Locations (1):
- People Science, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided